CLINICAL TRIAL: NCT05176587
Title: Medical and Medico-economic Evaluation Comparing the Follow-up of Patients Undergoing Bariatric Surgery (SPOC Study (Suivi Parcours Obésité en Chirurgie))
Brief Title: Medical and Medico-economic Evaluation Comparing the Follow-up of Patients Undergoing Bariatric Surgery
Acronym: SPOC
Status: Withdrawn | Type: Observational
Why Stopped: the deployment of the integrated pathwat takes longer than expected
Sponsor: Elsan (Other)
Collaborators: Cemka-Eval (Other)
Responsible Party: Sponsor
Other Study IDs: SPOC Study; 2021-A01847-34 (Other: ID-RCB)
Record Dates: First submitted 2021-12-21; First posted 2022-01-04 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Bariatric Surgery Candidate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Integrated group (SPOC)
  Interventions: Other: Follow-up of patients undergoing bariatric surgery : integrated pathway
- Control group

INTERVENTIONS:
Other: Follow-up of patients undergoing bariatric surgery : integrated pathway — Integrated pathway : multidisciplinary, pre- and post-operative, care course for patients undergoing bariatric surgery
  Groups: Integrated group (SPOC)

SUMMARY:
Study design :

Prospective, longitudinal, observational (non-interventional), multicenter, comparative medico-economic study - RIPH2, with direct matching to SNDS data (National Health Data System)

Main objective :

To evaluate the effectiveness of a multidisciplinary, pre- and post-operative, care course for patients undergoing bariatric surgery

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the Integrated group (SPOC)

  * Patient, male or female, at least 18 years old;
  * Patient undergoing bariatric surgery after the implementation of the integrated pathway (date depending on the deployment of the integrated pathway);
  * Patient informed and not objecting to this research;
  * Subject affiliated to or benefiting from a social security program.
* Inclusion criteria for the control group

  * Patient, male or female, at least 18 years old;
  * Patient undergoing bariatric surgery before the implementation of the integrated pathway (date depending on the deployment of the integrated pathway);
  * Patient informed and not objecting to this research;
  * Subject affiliated to or benefiting from a social security program.

Exclusion Criteria:

* • Protected patient : adult under tutorship, curatorship or other legal protection, deprived of his freedom by judiciary or administrative decision;

  * Patient hospitalised without consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Bariatric revision surgery at 5 years follow-up | 5 years after the first surgery
  Proportion of subjects who will have a bariatric revision surgery at 5 years follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- ELSAN, Paris, France

IPD SHARING:
Plan to Share IPD: No